CLINICAL TRIAL: NCT02661282
Title: A Phase I/II Clinical Trial of Autologous CMV-Specific Cytotoxic T Cells for GBM Patients
Brief Title: Autologous CMV-Specific Cytotoxic T Cells and Temozolomide in Treating Patients With Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0899; NCI-2016-00183 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0899 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-01-14; First posted 2016-01-22 (Estimated); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Cytomegalovirus Positive; Glioblastoma; Gliosarcoma; Malignant Glioma; Recurrent Brain Neoplasm; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (temozolomide, CMV-specific T cells, surgery) (Experimental): Patients receive temozolomide PO QD on days 1-21 and CMV-specific T cell transfer IV over 1-5 minutes on day 22. Patients undergo surgery on day 30 of cycle 1. Treatment repeats every 42 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive temozolomide PO QD on days 1-21. Treatment repeats every 42 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Autologous Cytomegalovirus-specific Cytotoxic T-lymphocytes; Other: Laboratory Biomarker Analysis; Drug: Temozolomide; Procedure: Therapeutic Conventional Surgery
- Arm II (temozolomide, CMV-specific T cells) (Active Comparator): Patients receive temozolomide PO QD on days 1-21 and CMV-specific T cell transfer intravenously IV over 1-5 minutes on day 22. Treatment repeats every 42 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Autologous Cytomegalovirus-specific Cytotoxic T-lymphocytes; Other: Laboratory Biomarker Analysis; Drug: Temozolomide; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Autologous Cytomegalovirus-specific Cytotoxic T-lymphocytes — Given IV
  Other Names: Autologous CMV-specific CTLs
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase I/II trial studies the side effects and best dose of autologous cytomegalovirus (CMV)-specific cytotoxic T cells when given together with temozolomide and to see how well they work in treating patients with glioblastoma. Autologous CMV-specific cytotoxic T cells may stimulate the immune system to attack specific tumor cells and stop them from growing or kill them. Drugs used in chemotherapy, such as temozolomide, may work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving autologous CMV-specific cytotoxic T cells with temozolomide may be a better treatment for patients with glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum feasible dose (MFD) or maximum tolerated dose (MTD) and safety of cytomegalovirus (CMV)-specific T cells in combination with dose-dense temozolomide in patients with recurrent glioblastoma. (Phase I) II. To evaluate the immunological effects in resected glioblastoma after intravenous administered cytomegalovirus (CMV)-stimulated adoptive T cells in patients with recurrent glioblastoma (GBM). (Phase II: recurrent glioblastoma undergoing resection) III. To correlate 6-month progression-free survival rate (PFS6) with objective clearance of CMV antigens as measured by immunohistochemistry (IHC) and by ex vivo T-cell-specific effector responses using intracellular cytokine profiling. (Phase II: recurrent glioblastoma undergoing resection) IV. Overall survival (OS). (Phase II: newly diagnosed glioblastoma)

SECONDARY OBJECTIVES:

I. Time to progression, overall survival (OS) as well as immunological reactivity and safety. (Phase II: recurrent glioblastoma undergoing resection) II. Safety and tolerability of dose-dense temozolomide in combination with intravenous administered CMV-stimulated adoptive T cells in patients receiving adjuvant therapy after completing external beam radiotherapy with concurrent temozolomide for newly diagnosed glioblastoma. (Phase II: newly diagnosed glioblastoma) III. Overall objective response rate (ORR), median duration of response, PFS6. (Phase II: newly diagnosed glioblastoma)

EXPLORATORY OBJECTIVES:

I. To determine the persistence and expansion of adoptively-infused CMV-specific T cells by multiparameter flow cytometry in serially-sampled peripheral blood. (Phase I) II. To identify imaging characteristics such as magnetic resonance imaging (MRI) textural analysis associated with immunological changes in tumor following treatment with CMV-stimulated adoptive T cells. (Phase II: recurrent glioblastoma undergoing resection) III. To ascertain if adoptive transfer of CMV-specific T cells leads to the expansion of T cells with specificity to other glioblastoma antigens (i.e. epitope spreading) by performing longitudinally monitoring of antigen-specific T cell frequency with enzyme-linked immunosorbent spot assay (ELISPOT). (Phase II: recurrent glioblastoma undergoing resection) IV. To determine the persistence and expansion of adoptively-infused CMV-specific T cells by multiparameter flow cytometry in serially-sampled peripheral blood. (Phase II: newly diagnosed glioblastoma)

OUTLINE: This is a phase I, dose-escalation study of CMV-specific T cells followed by a phase II study. Patients are assigned to 1 of 2 treatment arms.

ARM I: Patients receive temozolomide orally (PO) once a day (QD) on days 1-21 and CMV-specific T cell transfer intravenously (IV) over 1-5 minutes on day 22. Patients undergo surgery on day 30 of cycle 1. Treatment repeats every 42 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive temozolomide PO QD on days 1-21. Treatment repeats every 42 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive temozolomide PO QD on days 1-21 and CMV-specific T cell transfer intravenously IV over 1-5 minutes on day 22. Treatment repeats every 42 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial
* PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: Have histologically confirmed World Health Organization grade IV malignant glioma (glioblastoma or gliosarcoma); participants will also be eligible if the original histology was lower grade glioma and there is suspected transformation to glioblastoma based on imaging findings; if the final pathology report after resection fails to confirm recurrent glioblastoma or gliosarcoma, the subject will be followed for adverse events (AEs) and survival, but excluded for other primary and secondary objective analysis; the subject will be replaced
* PHASE II DOSE EXPANSION IN NEWLY DIAGNOSED GBM: Have histologically confirmed World Health Organization grade IV glioma (glioblastoma or gliosarcoma)
* PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: Be at first relapse; Note: relapse is defined as progression following initial therapy (i.e., radiation, chemotherapy, or radiation plus (+) chemotherapy); if the participant had a surgical resection for relapsed disease and no antitumor therapy instituted for up to 12 weeks, this is considered one relapse; for participants who had prior therapy for a lower grade glioma, the surgical diagnosis of glioblastoma or gliosarcoma will be considered first relapse
* PHASE II DOSE EXPANSION IN NEWLY DIAGNOSED GBM: Patients must have completed standard radiation therapy with concurrent temozolomide (TMZ) within 5 weeks (wks) of enrollment and must not have evidence of progressive disease on post treatment imaging; progression can only be defined using diagnostic imaging if there is new enhancement outside of the radiation field (beyond the high-dose region or 80% isodose line) or if there is unequivocal evidence of viable tumor on histopathologic sampling (e.g., solid tumor areas [i.e,> 70% tumor cell nuclei in areas], high or progressive increase in mindbomb homolog 1[MIB-1] proliferation index compared with prior biopsy, or evidence for histologic progression or increased anaplasia in tumor); Note: given the difficulty of differentiating true progression from pseudoprogression, clinical decline alone, in the absence of radiographic or histologic confirmation of progression, will not be sufficient for definition of progressive disease in the first 12 weeks after completion of concurrent chemoradiotherapy
* PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: Have measurable disease consisting of a minimal volume of 1 cm^3
* CMV seropositive
* PHASE I AND PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: Be willing to provide tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* PHASE II DOSE EXPANSION IN NEWLY DIAGNOSED GBM: Be willing to provide tissue from an archival tissue sample
* Have a performance status of >= 60 on the Karnofsky performance status (KPS)
* If patient is on steroids, patient must be on a stable or decreasing dose of steroids for 5 days, no more than 2 mg dexamethasone (or equivalent) total per day at the time of screening and consent; if on steroids at the time of screening, the dose will need to be tapered and discontinued at least 5 days prior to CMV T cell infusion
* Absolute neutrophil count (ANC) >= 1,500 /mcL (performed within 14 days [+3 working days] of treatment initiation)
* Platelets >= 100,000 / mcL (performed within 14 days [+3 working days] of treatment initiation)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (performed within 14 days [+3 working days] of treatment initiation)
* Serum creatinine OR measured or calculated (creatinine clearance should be calculated per institutional standard) creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 X upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (performed within 14 days [+3 working days] of treatment initiation)
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (performed within 14 days [+3 working days] of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X ULN (performed within 14 days [+3 working days] of treatment initiation)
* Coagulation international normalized ratio (INR) or prothrombin time (PT), activated partial thromboplastin time (aPTT) =< 1.5 X ULN (performed within 14 days [+3 working days] of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours of study enrollment; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control during the study and for 30 days after the last dose of the study drug or be surgically sterile; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception during the course of the study and for 30 days after the last dose of the study drug
* PHASE I: Have histologically confirmed World Health Organization WHO grade IV glioma (glioblastoma or gliosarcoma); participants will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of glioblastoma or variants is made
* PHASE I: A baseline brain MRI must be obtained no more than 14 days (+ 3 working days) prior to study enrollment; the patient must either be on no steroids or a stable dose of dexamethasone no greater than 2 mg a day for at least 5 days prior to entrance onto the study; patients having undergone recent surgery are eligible as long as they are at least 3 weeks from resection or 1 week from stereotactic biopsy, and recovering from any operative or perioperative complications; no measurable disease post resection will be required
* PHASE 1: Patients having undergone recent surgery are eligible as long as they are at least 3 weeks from resection or 1 week from stereotactic biopsy, and recovering from any operative or perioperative complications; no measurable disease post resection will be required
* PHASE I: Any number of prior relapses
* PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: A baseline brain MRI must be obtained no more than 14 days (+ 3 working days) prior to study enrollment; the patient must either be on no steroids or a stable dose of dexamethasone no greater than 2 mg a day for at least 5 days prior to entrance onto the study
* PHASE II DOSE EXPANSION IN NEWLY DIAGNOSED GBM: A baseline brain MRI obtained no more than 14 days (+ 3 working days) prior to study enrollment on a stable dose of steroids no greater than 2 mg a day of dexamethasone for at least 5 days, is required prior to entrance of a patient onto the study; patients must be registered on the study within 5 weeks of completion of concurrent chemoradiation

Exclusion Criteria:

* Has been treated previously with bevacizumab
* PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: Has tumor localized primarily to the posterior fossa, spinal cord, or an unresectable location
* Has received prior interstitial brachytherapy, implanted chemotherapy, or therapeutics delivered by local injection or convection enhanced delivery; prior treatment with Gliadel wafers will be excluded
* PHASE I AND PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: Is =< 12 weeks from completing external beam radiotherapy; patients with proven progressive disease (PD) by resection or with new lesions outside of the radiation field should not be excluded even if they are within 12 weeks of external radiation therapy (XRT), per Response Assessment in Neuro-Oncology (RANO) criteria for early PD
* PHASE I AND PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: Is currently participating in a study of an investigational agent or using an investigational device for therapeutic purposes; concurrent use of Optune device is not allowed
* PHASE II DOSE EXPANSION IN NEWLY DIAGNOSED GBM: Is currently participating or has participated in any other newly diagnosed therapeutic trial before or after chemoradiation
* CMV seronegative
* Has a known history of human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies); human T-cell lymphotropic virus (HTLV) 1 antibody (HTLV1) and/or HTLV2; active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected); patients with prior hepatitis B virus (HBV) vaccination (anti-hepatitis B surface antibody [HBs] positive, HBsAg negative, anti-hepatitis B core antibody [HBc] negative) will NOT be excluded
* Has a diagnosis of immunodeficiency or is receiving systemic immunosuppressive therapy within 7 days of study entrance
* PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: Has had prior chemotherapy, or targeted small molecule therapy, within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent; Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study; Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: Has known gliomatous meningitis, subependymal spread, extracranial disease, or multifocal disease
* PHASE II DOSE EXPANSION IN NEWLY DIAGNOSED GBM: Has known gliomatous meningitis, extracranial disease, or multifocal disease
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit
* PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION AND IN NEWLY DIAGNOSED GBM: Has received prior therapy with any antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Contraindication for undergoing MRIs
* PHASE II DOSE EXPANSION IN RECURRENT GBM UNDERGOING RESECTION: Evidence of bleeding diathesis or use of anticoagulant medication or any medication that may increase the risk of bleeding that cannot be stopped prior to surgery
* PHASE I: Tumor localized primarily to the posterior fossa or spinal cord
* PHASE I: Has known gliomatous meningitis, subependymal spread, or extracranial disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shiao-Pei Weathers, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I/II CMV Clinical trial TCELL ( Leukapheresis performed over2-3 hrs to collect white blood cells. Will start receiving Temozolomide and CMV CTLs
Pre-assignment Details: 65 participants were consented, 40 participants were inevaluable
Groups:
- Phase I: Recurrent Glioblastoma Dose Level 5 x 10^6; Phase I: Recurrent Glioblastoma Dose Level 1 x 10^7; Phase I: Recurrent Glioblastoma Dose Level 5 x 10^7; Phase I: Recurrent Glioblastoma Dose Level 1 x 10^8: Dose escalation component in participants with recurrent glioblastoma to determine the maximum feasible dose (MFD) or maximum tolerated dose (MTD) of CMV-specific T cells in combination with dose-dense temozolomide. We will follow a 3+3 design exploring 4 dose levels of CMV-T cells: 5 x 106, 1 x 107, 5 x 107, and 1 x 108 CMV CTLs. 4 cycles total of dose-dense TMZ and CMV-T cell infusion. Following completion of 4 cycles of dose-dense TMZ and CMV-T cell infusion, participants can receive additional 42-day cycles of dose-dense TMZ for up to 12 cycles or tumor PD.
- Phase II: Newly Diagnosed Dose Level 1 x 10^8: Participants will receive 4 cycles total of dose-dense TMZ followed by adoptive CMV T cell infusion. Following completion of 4 cycles of dose-dense TMZ and CMV T cell infusion, patients can receive standard dose TMZ 200 mg/m^ 2 days 1-5 every 28 days up to 12 cycles or tumor PD.
- Phase II: Recurrent Glioblastoma Dose Level 1 x 10^8: Participants will receive a total of 3 cycles of dose-dense temozolomide followed by fixed doses of CMV-specific T cell infusion in the post-surgical phase, after which they can remain on dose-dense temozolomide until tumor progression, as long as there are no unacceptable toxicities or until completion of 12 cycles of treatment with dose-dense temozolomide (whichever occurs first).
Period: Overall Study
Arm/Group | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^6 | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^7 | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^7 | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^8 | Phase II: Newly Diagnosed Dose Level 1 x 10^8 | Phase II: Recurrent Glioblastoma Dose Level 1 x 10^8
Started | 3 | 3 | 3 | 7 | 3 | 1
Completed | 3 | 3 | 3 | 7 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II: Newly Diagnosed Dose Level 1 x 10^8: Participants received 4 cycles total of dose-dense TMZ followed by adoptive CMV T cell infusion. Following completion of 4 cycles of dose-dense TMZ and CMV T cell infusion, patients can receive standard dose TMZ 200 mg/m^ 2 days 1-5 every 28 days up to 12 cycles or tumor PD.
- Total: Total of all reporting groups
Arm/Group | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^6 | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^7 | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^7 | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^8 | Phase II: Newly Diagnosed Dose Level 1 x 10^8 | Phase II: Recurrent Glioblastoma Dose Level 1 x 10^8 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 3 | 1 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 6 | 3 | 1 | 19
  >=65 years | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 4 | 1 | 0 | 10
  Male | 0 | 3 | 1 | 3 | 2 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 2 | 2 | 2 | 7 | 3 | 1 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 3 | 7 | 3 | 1 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 7 | 3 | 1 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Recurrent Glioblastoma Participant Cohort)- Phase I
Description: The number of participants who were treated at the respective dose level without DLT
Time Frame: Up to 42 days
Measure: Number; unit: participants
Groups:
- Phase I: Recurrent Glioblastoma (MTD) Dose Level 1 x 10^8: Dose escalation component in participants with recurrent glioblastoma to determine the maximum feasible dose (MFD) or maximum tolerated dose (MTD) of CMV-specific T cells in combination with dose-dense temozolomide. We will follow a 3+3 design exploring 4 dose levels of CMV-T cells: 5 x 106, 1 x 107, 5 x 107, and 1 x 108 CMV CTLs. 4 cycles total of dose-dense TMZ and CMV-T cell infusion. Following completion of 4 cycles of dose-dense TMZ and CMV-T cell infusion, participants can receive additional 42-day cycles of dose-dense TMZ for up to 12 cycles or tumor PD.
Arm/Group | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^6 | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^7 | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^7 | Phase I: Recurrent Glioblastoma (MTD) Dose Level 1 x 10^8
Number analyzed (Participants) | 3 | 3 | 3 | 7
participants | 3 | 3 | 3 | 7

2. Primary Outcome: Number of Participants With Immunological Effects in Tumor Tissue (Recurrent Glioblastoma Cohort)- Phase II
Description: Descriptive statistics will be used to summarize immunological effect. To evaluate the tumor-mediated immune suppression at the effector location, the markers (interferon, interleukin-2, and tumor necrosis factor alpha, perforin, granzyme B) will be measured for immune responses in the tumor microenvironment rather than in the peripheral blood.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: Recurrent Glioblastoma Dose Level 1 x 10^8: Participants will receive a total of 3 cycles of dose-dense temozolomide (TMZ) followed by fixed doses of CMV-specific T cell infusion in the post-surgical phase, after which they can remain on dose-dense temozolomide until tumor progression, as long as there are no unacceptable toxicities or until completion of 12 cycles of treatment with dose-dense temozolomide (whichever occurs first).
Arm/Group | Phase II: Recurrent Glioblastoma Dose Level 1 x 10^8
Number analyzed (Participants) | 1
Participants | 1

3. Primary Outcome: Progression Free Survival (PFS) (Recurrent Glioblastoma Cohort) at 6 Months- Phase II
Description: Progression-free survival (PFS) is defined as the time from study enrollment until the time of first disease progression, relapse, or death due to disease. Patients who are alive without progression or relapse will be censored at the time of last contact. The point estimate of 6-month progression-free survival (PFS6) will be analyzed. Kaplan-Meier curves will be generated and median survival time will be derived.
Time Frame: 6 months
Measure: Number; unit: months
Arm/Group | Phase II: Recurrent Glioblastoma Dose Level 1 x 10^8
Number analyzed (Participants) | 1
months | 2.5

4. Primary Outcome: Overall Survival (OS) (Newly Diagnosed Glioblastoma Cohort)- Phase II
Description: Overall Survival is defined as the time from definitive histological diagnosis until the time of death.
Time Frame: Time from definitive histological diagnosis until death
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase II: Newly Diagnosed Dose Level 1 x 10^8
Number analyzed (Participants) | 3
weeks | 24 [13 to 24]

5. Secondary Outcome: Time to Progression (Recurrent Glioblastoma Cohort)- Phase II
Description: The length of time from the date of diagnosis or the start of treatment for a disease until the disease starts to get worse or spread to other parts of the body.
Time Frame: Baseline to disease progression, assessed up to 4 years
Measure: Number; unit: months
Arm/Group | Phase II: Recurrent Glioblastoma Dose Level 1 x 10^8
Number analyzed (Participants) | 1
months | 2.5

6. Secondary Outcome: Overall Objective Response Rate (ORR) (Newly Diagnosed Glioblastoma Cohort)- Phase II
Description: The number of participants with stable disease according to Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Newly Diagnosed Dose Level 1 x 10^8
Number analyzed (Participants) | 3
Participants | 3

7. Secondary Outcome: Median Duration of Response (Newly Diagnosed Glioblastoma Cohort)- Phase II
Description: Cox proportional hazard regression will be employed for multivariate analysis.
Time Frame: Baseline to response, assessed up to 4 years
Measure: Median (Full Range); unit: months
Arm/Group | Phase II: Newly Diagnosed Dose Level 1 x 10^8
Number analyzed (Participants) | 3
months | 5.3 [4 to 10]

8. Secondary Outcome: Progression Free Survival (PFS) (Newly Diagnosed Glioblastoma Cohort)- Phase II
Description: Progression free survival is defined as time in weeks from start of study treatment to first documentation of objective tumor progression or up to death due to any cause, whichever occurs first.
Time Frame: At 6 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase II: Newly Diagnosed Dose Level 1 x 10^8
Number analyzed (Participants) | 3
weeks | 19 [9 to 20]

ADVERSE EVENTS:
Time Frame: from the first dose through 30 days after the completion of study treatment, up to 4 years
Description: No Phase 2 participants died and 13 out of 16 Phase 1 participants died unrelated to study treatment. For the Phase 2 newly diagnosed participants the median survival weeks was 24 at the time of last follow up.
Arm/Group | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^6 | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^7 | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^7 | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^8 | Phase II: Newly Diagnosed Dose Level 1 x 10^8 | Phase II: Recurrent Glioblastoma Dose Level 1 x 10^8
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/3 | 3/3 | 7/7 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/3 | 3/7 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/3 | 5/7 | 2/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^6 (N=3) | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^7 (N=3) | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^7 (N=3) | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^8 (N=7) | Phase II: Newly Diagnosed Dose Level 1 x 10^8 (N=3) | Phase II: Recurrent Glioblastoma Dose Level 1 x 10^8 (N=1)
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Surgical and medical procedures, other-removal of facial cyst (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cognitive Disturbance (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^6 (N=3) | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^7 (N=3) | Phase I: Recurrent Glioblastoma Dose Level 5 x 10^7 (N=3) | Phase I: Recurrent Glioblastoma Dose Level 1 x 10^8 (N=7) | Phase II: Newly Diagnosed Dose Level 1 x 10^8 (N=3) | Phase II: Recurrent Glioblastoma Dose Level 1 x 10^8 (N=1)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Cognitive Disturbance (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 2 | 4 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Malaise (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Nausea (General disorders) | 0 | 3 | 0 | 0 | 0 | 0
Fatigue (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Weight loss (Investigations) | 3 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1 | 1 | 2 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 1 | 0
Concentration impairment (Nervous system disorders) | 1 | 1 | 1 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 2 | 2 | 1 | 3 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Decreased platelet count (Investigations) | 0 | 1 | 0 | 2 | 0 | 0
Decreased lymphocyte count (Investigations) | 0 | 2 | 1 | 2 | 0 | 0
Decreased neutrophil count (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT02661282/Prot_SAP_000.pdf